CLINICAL TRIAL: NCT05262114
Title: Would You be Happy to be Contacted About Research?
Acronym: The Who
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0322-21; IRAS Number: 291348 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2021-11-25; First posted 2022-03-02 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Patient Acceptability to Being Invited to Take Part in Research of Relevance to Them

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-cursor text: A pre-notification text message (SMS) will be sent to eligible people informing them of their imminent invitation to participate in The Who, two days later a brief text message (SMS) will be sent from the general practice to eligible people, inviting them to participate in The Who.
- Invitation only: A brief text message (SMS) will be sent from the general practice to eligible people, inviting them to participate in The Who.

SUMMARY:
The aim of this study is to re-examine the proportion of primary care patients that would be happy to be contacted about research of relevance to them. This study will examine the utility of SMS messages sent to patients by their general practice, with a link URL to an online questionnaire containing five research questions.

DETAILED DESCRIPTION:
Since the onset of the COVID-19 pandemic in 2019, the NIHR has played a critical role in the fight against this new disease with the delivery of COVID-19 research studies. Taking part in COVID-19 research is vital to enable effective treatments to be identified, evidenced and made available to NHS patients as quickly as possible. Over 100,000 UK participants have now enrolled in COVID-19 urgent public health research supported by the NIHR.

Keele Clinical Trials Unit (CTU) quickly implemented online data collection methodologies during 2020, in order to continue with recruitment of and retention of research participants and in response to the national lockdown and tiered systems implemented for protection of the population during the pandemic. There is now opportunity, to re-evaluate the proportion of primary care patients that would be happy to be contacted about research of relevance and also to assess the utility of online technologies, in particular SMS text messaging and an online survey platform, in the collection of the research data.

The specific research objectives of this study are:

1. To examine patient response rates to an invitation to complete an online Keele Health Survey questionnaire, delivered by SMS message from their general practice,
2. To examine the difference in patient response rates to the invitation to participate in the research study with and without a precursor test message (SMS).
3. To estimate the number of patients that would be happy to be contacted about future research studies relevant to their health.
4. To explore any demographic variances in completion responses.
5. To estimate research question completion rate feasibility, for future use of SMS messages containing a link URL to an online Keele Health Survey questionnaire to collect research data.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years or over
* Mobile telephone number must be registered at general practice (doctor's surgery)

Exclusion Criteria:

* Anyone under the age of 18
* Anyone who does not have their mobile phone number registered with their general practice (doctor's surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of individuals who are aged 18 years of age or older and must have their mobile phone number registered with their general practice. Participants will be registered with a GP surgery within the West Midlands CRN network of practices, situated within England, UK.
Sampling Method: Non-Probability Sample
Enrollment: 20969 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Estimate the proportion of people happy to be contacted by their practice | Over 4 weeks
  To estimate the proportion of people who are happy for their practice to contact them about any future research studies, which are relevant to their health.

SECONDARY OUTCOMES:
Patient response rates to invitation | Over 4 weeks
  To examine patient response rates to an invitation to complete an online questionnaire, delivered by SMS message from their general practice,
Examine response rates using a precursor text message | Over 4 weeks
  To examine the difference in patient response rates to the invitation to participate in the research study with and without a precursor test message (SMS).
Explore any demographic variances in completion responses. | Over 4 weeks
  Compare self reported data. age, gender, ethnicity,
To estimate research question completion rate feasibility | Over 4 weeks
  Estimationg the completion rates of the questionnaires will help to inform the future use of SMS messages and online questionnaires to collect research data.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lawton, MPhil, Principal Investigator — Head of Operations - Clinical Trials Unit; Christian Mallen, Professor, Study Director — Head of School of Medicine
Locations (1):
- Keele University: School of Medicine, Newcastle-under-Lyme, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No